CLINICAL TRIAL: NCT02189629
Title: A LONG-TERM SAFETY AND EFFICACY STUDY OF CD5789 (Trifarotene) 50 µg/g CREAM IN SUBJECTS WITH ACNE VULGARIS
Brief Title: CD5789 (Trifarotene) Long Term Safety Study on Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06.SPR.18250
Record Dates: First submitted 2014-07-11; First posted 2014-07-14 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Acne Vulgaris
Keywords: Acne vulgaris; Safety; Face; Trunk
MeSH Terms: conditions — Acne Vulgaris; Facies | interventions — trifarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD5789 (trifarotene) cream (Experimental)
  Interventions: Drug: CD5789 (trifarotene)

INTERVENTIONS:
Drug: CD5789 (trifarotene)

SUMMARY:
Multi-center, open-label, non-comparative safety and efficacy study with 52 Weeks of treatment on the face and trunk for acne vulgaris.

DETAILED DESCRIPTION:
To determine the safety and efficacy of CD5789 (trifarotene) 50 µg/g cream in the long-term treatment (up to 52 Weeks) of subjects with acne vulgaris. Efficacy will be evaluated as a secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* The Subject has a facial acne severity grade of IGA grade 3 (moderate) at Screening and Baseline visits.
* The Subject has a minimum of 20 inflammatory lesions and 25 non-inflammatory lesions at Screening and Baseline visits on the face.
* Exclusion Criteria:
* The subject has severe forms of acne (acne conglobata, acne fulminans) or secondary acne form (chloracne, drug-induced acne, etc.).
* The Subject has more than 1 nodule on the face at Screening and at Baseline visits.
* The Subject has any acne cyst on the face at Screening and at Baseline visits.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Chan, Study Director — Galderma R&D
Locations (31):
- United States (14):
  - Galderma Investigational Site, Mobile, Alabama
  - Galderma Investigational Site, Rogers, Arkansas
  - Galderma Investigational Site, Sacramento, California
  - Galderma Investigational Site, San Diego, California
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, Miramar, Florida
  - Galderma Investigational Site, Newnan, Georgia
  - Galderma Investigational Site, Louisville, Kentucky
  - Galderma Investigational Site, Albuquerque, New Mexico
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational Site, High Point, North Carolina
  - Galderma Investigational Site, Beachwood, Ohio
  - Galderma Investigational Site, Portland, Oregon
  - Galderma Investigational Site, Knoxville, Tennessee
- Czechia (5):
  - Galderma Investigational Site, Chomutov
  - Galderma Investigational site, Hradec Králové
  - Galderma Investigational Site, Olomouc
  - Galderma Investigational Site, Pardubice
  - Galderma Investigational site, Prague
- Germany (6):
  - Galderma Investigational Site, Augsburg
  - Galderma Investigational Site, Berlin
  - Galderma Investigational Site, Dessau
  - Galderma Investigational Site, Mahlow
  - Galderma Investigational Site, Münster
  - Galderma Investigational Site, Wuppertal
- Hungary (6):
  - Galderma Investigational Site, Balatonfüred
  - Galderma Investigational Site, Miskolc
  - Galderma Investigational Site, Pécel
  - Galderma Investigational Site, Szeged
  - Galderma Investigational Site, Szekszárd
  - Galderma Investigational Site, Szolnok

RESULTS

PARTICIPANT FLOW:
Groups:
- CD5789 Cream: CD5789 Trifarotene 50 microgram/gram cream
Period: Overall Study
Arm/Group | CD5789 Cream
Started | 453
Completed | 348
Not Completed | 105

BASELINE CHARACTERISTICS:
Population: A total of 455 subjects were enrolled and 453 were exposed to CD5789 50 microgram/gram cream for up to 52 weeks.
Groups:
- CD5789 Cream: CD5789 Trifarotene 50 microgram/gram
Arm/Group | CD5789 Cream
Number analyzed (Participants) | 453
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 286
  Between 18 and 65 years | 167
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 226
  Male | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47
  Not Hispanic or Latino | 406
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 12
  White | 432
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 91
  United States | 163
  Czechia | 104
  Germany | 95

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) Success Rate up to Week 52
Description: Number of subjects who achieved an Investigator Global Assessment (IGA) score of 1 (almost clear) or 0 (clear).
Time Frame: From Baseline to Week 52
Population: A total of 455 subjects were enrolled in the study, of whom 453 were treated with CD5789 50 microgram/gram.
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 Cream
Number analyzed (Participants) | 453
Participants | 453

2. Secondary Outcome: Physician Global Assessment (PGA) Success Rate up to Week 52
Description: Number of subjects who achieved a Physician Global Assessment (PGA) score of 1 (almost clear) or 0 (clear).
Time Frame: From Baseline to Week 52
Population: A total of 455 subjects were enrolled in the study, of whom 453 were treated with CD5789 50 microgram/gram
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 Cream
Number analyzed (Participants) | 453
Participants | 453

ADVERSE EVENTS:
Time Frame: Over 52 Weeks
Arm/Group | CD5789 Cream
All-Cause Mortality (participants affected / at risk) | 0/453
Serious Adverse Events (participants affected / at risk) | 10/453
Other Adverse Events (participants affected / at risk) | 170/453
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 Cream (N=453)
Crohn's Disease (Gastrointestinal disorders) | 1
Umbilical Hernia (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 1
Complex partial seizures (Nervous system disorders) | 1
Complex regional Pain syndrome (Nervous system disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Liver function test abnormal (Investigations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 Cream (N=453)
Sunburn (Injury, poisoning and procedural complications) | 27
Ligament Sprain (Injury, poisoning and procedural complications) | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 9
Headache (Nervous system disorders) | 6
Application Site Pruritis (General disorders) | 23
Application Site Irritation (General disorders) | 22
Diarrhea (Gastrointestinal disorders) | 5
Acne (Skin and subcutaneous tissue disorders) | 5
Nasopharyngitis (Infections and infestations) | 48
Upper Respiratory Tract Infection (Infections and infestations) | 13
Influenza (Infections and infestations) | 9
Infectious Mononucleosis (Infections and infestations) | 5
Tonsillitis (Infections and infestations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data or results arising out of the study will not be presented or published in any form or media by the PI/Institution without the prior written consent of sponsor.

DOCUMENTS (2):
  • Study Protocol (2014-08-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT02189629/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT02189629/SAP_002.pdf